CLINICAL TRIAL: NCT04560959
Title: An Atlas of Cerebral Responses to the Stimuli of the tACS Recorded by SEEG
Brief Title: Atlas of Intracranial Recordings on Cortical Responses After Functional tACS
Acronym: AIRCRAFT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYS-[2020]-051
Record Dates: First submitted 2020-08-07; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-08

CONDITIONS: Transcranial Alternating Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- tACS arm (Experimental): The patient would receive strings of tACS stimulations in 77.5 HZ, each string would last for 1 second, followed by an interval of 5 seconds. A total of 600 strings would be sent out to the patients.
  Interventions: Device: tACS

INTERVENTIONS:
Device: tACS — tACS would be performed to epilepsy patients who have already received implantation of the SEEG electrodes

SUMMARY:
By analyzing the SEEG recordings, we explore the range of cortical functional responses to strings of 77.5Hz stimulations delivered by tACS,

ELIGIBILITY:
Inclusion Criteria:

* All epileptic patients that would receive the implantation of SEEG electrodes, regardless of the seizure locations;
* There was no metal implantation before;
* Eligible for MRI examination;
* No other lesional neurological disorders;
* Could be well informed by the study protocols.

Exclusion Criteria:

* Suffered from any other mental illnesses prior to the enrollment;
* Those suffering from the serious or unstable organic diseases;
* Pregnant or lactation women, and those who have a plan of pregnant;
* Patients with central nervous system tumors, acute brain injury or infection;
* Skin injured, or allergic to the exposure of the conductive gel;
* Those with implanted devices;
* Those who received modified electrical convulsive therapy, or TMS within the recent one month;
* The score of item 3 (suicidal item) in HAMD-17 equal or greater than 3;
* Enrolled in any other on going trials;
* Other situations evaluated by the researchers as inappropriate to the enrollment

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-20 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes of intracranial activities | Within 250 ms immediately after the stimulation.
  The change of the power in a band of 0-200 HZ according to the intracranial EEG recording.

SECONDARY OUTCOMES:
Frequency of the epileptic discharges | 50 minutes during the stimulation and 50 minutes of the interictal baseline before the intervention during the same hour of the day
  To count the numbers of epileptic discharges within the same duration before and when tACS intervention.
Event related potential (ERP) | Baseline: 24 hours before the tACS intervention; Observation: Immediately after the end of the tACS intervention.
  ERP related to cognitive tasks before and immediately after the tACS intervention

CONTACTS AND LOCATIONS:
Overall Officials: G.G. Zhao, Principal Investigator — Department of Neurosurgery, Capital Medical University

REFERENCES:
- [Derived] Shan Y, Wang H, Yang Y, Wang J, Zhao W, Huang Y, Wang H, Han B, Pan N, Jin X, Fan X, Liu Y, Wang J, Wang C, Zhang H, Chen S, Liu T, Yan T, Si T, Yin L, Li X, Cosci F, Zhang X, Zhang G, Gao K, Zhao G. Evidence of a large current of transcranial alternating current stimulation directly to deep brain regions. Mol Psychiatry. 2023 Dec;28(12):5402-5410. doi: 10.1038/s41380-023-02150-8. Epub 2023 Jul 19. PMID 37468529